CLINICAL TRIAL: NCT01414036
Title: Primary Care-based Patient Navigation to Promote Smoking Cessation Treatment: a Pilot Randomized Controlled Trial
Brief Title: Pilot Study of Patient Navigation to Promote Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Karen E. Lasser, Physician, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UL1RR025771 (NIH); UL1RR025771 (NIH)
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Cigarette Smoking
Keywords: cigarette smoking; patient navigation; primary care
MeSH Terms: conditions — Cigarette Smoking | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Traditional Care control (Active Comparator): This arm will receive a low literacy smoking cessation educational brochure, a list of hospital and community resources for smoking cessation, in addition to usual care.
  Interventions: Other: Enhanced Traditional Care control
- Patient Navigation (Experimental): Patients in this arm will receive a low literacy smoking cessation educational brochure and a list of hospital and community resources for smoking cessation. Patients will also receive navigation from a trained navigator Patients will receive up to 4 hours of patient navigation, in person or over the phone, over a 3-month period.
  Interventions: Behavioral: Patient navigation

INTERVENTIONS:
Other: Enhanced Traditional Care control — Educational brochure, list of hospital and community resources
  Arms: Enhanced Traditional Care control
Behavioral: Patient navigation — Patients will receive up to 4 hours of patient navigation, in person or over the phone, over a 3-month period.
  Arms: Patient Navigation

SUMMARY:
Cigarette smoking is a highly significant health threat, responsible for more than 430,000 deaths each year. Low-income persons and racial/ethnic minorities are at particularly high risk, smoking at greater rates and having greater tobacco-related morbidity and mortality than other persons. Yet poor and minority smokers are less likely to receive advice to stop smoking or to use tobacco cessation services. Using non-physician members of the health care team as patient navigators to connect low-income and minority smokers to evidence-based tobacco treatment services is a promising approach because 1) many primary care providers (PCPs) are unable to provide counseling to patients who smoke due to time constraints; 2) minority patients may be less aware of smoking cessation resources and may have misconceptions about tobacco dependence treatments; and 3) as primary care practices are redesigned as medical homes, non-physician members of the health care team will increasingly be taking on tasks previously performed by PCPs. Patient navigators are lay persons from the community, working as paid employees, who are trained to guide patients through the health care system to receive services. Information on the efficacy of patient navigation to connect vulnerable patients to smoking cessation services is needed.

The investigators will implement a patient navigation-based intervention in the primary care setting to promote engagement of low-income and minority patients in smoking cessation treatment. To test our intervention, the investigators will conduct a pilot randomized control trial (RCT), randomizing 240 patients to the intervention condition (patient navigation) or an enhanced traditional care (ETC) control condition. The investigators will perform follow-up at three months following the start of the intervention, with a primary outcome of engagement in smoking cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years
2. smoked cigarettes in the past week
3. have a scheduled visit with a PCP
4. telephone access
5. English speaking
6. able and willing to participate in the study protocol and provide informed consent.

Exclusion Criteria:

1. planning to move out of the area within the next 6 months
2. cognitive impairments that preclude participation in study activities.
3. severe illness or distress
4. inability to read/understand English
5. actively using evidence-based smoking cessation treatment, and
6. transient residence or lack of a telephone for follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Lasser, MD, MPH, Principal Investigator — Boston Medical Center/Boston University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
J Ethn Subst Abuse. 2013 ; 12(4): . doi:10.1080/15332640.2013.819311.
  http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3827692/

RESULTS

PARTICIPANT FLOW:
Period: Received Allocated Intervention
Arm/Group | Enhanced Traditional Care Control | Patient Navigation
Started | 23 | 24
Completed | 23 | 11
Not Completed | 0 | 13
Period: Completed 3 Month Survey
Arm/Group | Enhanced Traditional Care Control | Patient Navigation
Started | 23 | 24
Completed | 14 | 19
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Traditional Care Control | Patient Navigation | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 47
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Engagement in Smoking Cessation Treatment
Description: This is a dichotomous variable, Y/N, based on a) completion of > 1 quit line counseling session (based on self-report) OR b) > 1 PCP visit in which smoking cessation treatment is discussed (patient self-report and medical record review of progress notes) OR c) Completion of > 1 session of a BMC smoking cessation group (medical record review).
Time Frame: 3 months
Population: 14 out of the 23 in control group completed 3 month survey and 19 out of 24 in patient navigation group completed the 3 month survey.
Measure: Number; unit: participant
Arm/Group | Enhanced Traditional Care Control | Patient Navigation
Number analyzed (Participants) | 14 | 19
participant | 7 | 9

2. Secondary Outcome: Stage of Change With Regard to Smoking Cessation
Description: Stage of change is assessed at baseline and 3 months. Three months after study entry, 7 of patient navigation-intervention participants who had initially said that they did not have a time frame in mind for quitting reported that they now had a time frame in mind for quitting, relative to 1 of ETC-control participants.
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Enhanced Traditional Care Control | Patient Navigation
Number analyzed (Participants) | 14 | 19
participant | 1 | 7

3. Secondary Outcome: Use of Other Tobacco Treatment Support
Description: self-report of all tobacco treatment support received, including support from non-study sources, including the internet, during the study period.
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Enhanced Traditional Care Control | Patient Navigation
Number analyzed (Participants) | 14 | 19
participant | 6 | 9

ADVERSE EVENTS:
Arm/Group | Enhanced Traditional Care Control | Patient Navigation
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No